CLINICAL TRIAL: NCT02512887
Title: Caudal vs Local Anesthesia in Hypospadias: The CLASH Study
Brief Title: Caudal vs Local Anesthesia in Hypospadias
Acronym: CLASH
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: McMaster University (Other)
Collaborators: Canadian Urological Association (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CLASH
Record Dates: First submitted 2015-07-27; First posted 2015-07-31 (Estimated); Last update posted 2023-03-15 (Actual); Status verified 2023-03

CONDITIONS: Hypospadias
Keywords: Hypospadias; Caudal Block; Dorsal Penile Block; Anesthesia; Complications; Post-operative; Urethrocutaneous Fistula; Glans dehiscence
MeSH Terms: conditions — Hypospadias | interventions — Anesthesia, Local

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Caudal Block Anesthesia (Experimental): Anesthesia will be delivered via inhalation induction with air/nitrous oxide and sevoflurane, and injection of 0.25% bupivacaine 1mL/kg without epinephrine into the caudal canal, which is the sacral portion of the spinal canal.
  Interventions: Drug: Caudal Block Anesthesia
- Dorsal Penile Block Anesthesia (Active Comparator): Anesthesia will be delivered via inhalation induction with air/nitrous oxide and sevoflurane, and injection of 0.25% bupivacaine without epinephrine into the dorsal portion of the penis.
  Interventions: Drug: Dorsal Penile Block Anesthesia

INTERVENTIONS:
Drug: Caudal Block Anesthesia — Anesthesia will be delivered via inhalation induction with air/nitrous oxide and sevoflurane, and injection of 0.25% bupivacaine 1mL/kg without epinephrine into the caudal canal, which is the sacral portion of the spinal canal.
  Arms: Caudal Block Anesthesia
Drug: Dorsal Penile Block Anesthesia — Anesthesia will be delivered via inhalation induction with air/nitrous oxide and sevoflurane, and injection of 0.25% bupivacaine without epinephrine into the dorsal portion of the penis.
  Other Names: Local Anesthesia
  Arms: Dorsal Penile Block Anesthesia

SUMMARY:
Hypospadias is one of the most common congenital malformations of the genitalia in boys, and is typically managed by surgical intervention. During pediatric urological surgery, caudal anesthesia is one of the most common regional anesthetic techniques used. Also known as caudal block, it has been shown to be a safe and effective anesthetic technique in children with a low incidence of anesthesia-related complications.While the reported incidence of complications directly associated with caudal block is low, there is scarce and inconclusive evidence on the impact of caudal anesthesia on the incidence of surgical complications. As a result, the objective of this superiority, randomized controlled trial is to assess whether the use of caudal anesthesia, when compared to dorsal penile block, is associated with a higher rate of urethrocutaneous fistulas and glans dehiscence post hypospadias repair.

DETAILED DESCRIPTION:
The rationale to conduct a definitive study comes as a result of the limitations inherent in the pre-existing literature due to selection bias, and the primarily retrospective nature of the current evidence, which is unclear whether caudal blocks result in higher complication rates following hypospadias repair. The only way to close this knowledge gap and disturb the current state of clinical equipoise surrounding this topic is to randomly assign the two interventions (caudal or penile block) to patients undergoing hypospadias repair. The rationale to conduct this pilot study is to determine whether the definitive study is feasible and to ensure that any methodological issues are identified and addressed prior to investing significant resources in a definitive trial.

This study will be a pilot study to determine the feasibility of conducting a large definitive superiority, parallel, randomized controlled trial (RCT) to assess whether dorsal penile block results in fewer postoperative complications than caudal block in boys (6-48 mos.) undergoing hypospadias repair.

Hypospadias repair will be carried out under standardized analgesic administration.. Participants may be given fentanyl (1-3 mcg/kg) at the discretion of the anesthesiologist. Anesthesia will be delivered to all participants via inhalation induction with air/nitrous oxide and sevoflurane. In addition either caudal anesthetic block (0.25% bupivacaine 1 ml/kg to a maximum of 10 ml) or dorsal penile block (bupivacaine without epinephrine 10-20 ml/kg) will be administered based on our randomization scheme. Each patient will also receive antiemetic prophylaxis with dexamethasone 150 mcg/kg ondansetron 50 mcg/kg Acetaminophen suppository 40 mg/kg, and intravenous morphine (0.02-0.1 mg/kg).

At Home At home, Oral Morphine (0.2 mg/kg) q4h prn, Ditropan (0.2 mg/kg) q12h prn, Tylenol (15 mg/kg/dose) q4h or Ibuprofen (10 mg/kg/dose) q6h will be prescribed at discharge to be administered at the parents' discretion. Trimethoprim (2 mg/kg) will also be prescribed for administration until catheter removal.

ELIGIBILITY:
Inclusion Criteria:

* Males 6-48 months of age at presentation to Pediatric Urology clinics
* Patient who requires hypospadias repair by fellowship-trained Pediatric Urologists.

Exclusion Criteria:

* Patients who have undergone previous hypospadias surgery
* Patients who have contraindications to either caudal or dorsal penile block
* Inability of parent/guardian to understand English/French
* Deviation to pre-established anesthesia protocol

Ages: 6 Months to 48 Months | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 224 (Estimated)
Dates: Start 2016-07; Primary Completion 2024-01 (Estimated); Study Completion 2024-01 (Estimated)

PRIMARY OUTCOMES:
Post-operative Complication Rate | Follow-up to assess the complications, specifically urethrocutaneous fistula (UCF) and glans dehiscence within 12 months post-surgery.
  UCF is defined as an abnormal communication between the reconstructed urethra and the skin located between the original meatus and the tip of the penis.Glans dehiscence is considered as a complete separation of the glans wings with or without a band of skin between them.
Recruitment rate | trial duration 1 year
  Percentage of eligible participants enrolled, Randomization rate (percentage of enrolled participants randomized)
Protocol violations or Adverse events | trial duration 1 year
  Frequency of protocol violations or adverse events related to the study intervention.

SECONDARY OUTCOMES:
Operating Room (OR) time | Record duration of operative time (takes on average 30-45 minutes)
  OR time will be measured in minutes from the time the patient enters the OR to the time surgery is complete
Complications directly related to caudal block | Complications will be measured at a clinic visit 48 hours after surgery.
  Complications directly related to caudal block include block failure, blood aspiration and intravascular injections.
Complications directly related to dorsal penile block | Complications will be measured at a clinic visit 48 hours after surgery.
  Complications directly related to dorsal penile block include hematoma and intravascular injection.
Post-operative Pain | Measure at patient admission and discharge at 30 minute intervals.
  Pain scores will be measured through a reliable and validated observer-rated Face, Legs, Activity, Cry, Consolability (FLACC) Behavioural Scale by two trained, blinded, and independent study personnel. Both study personnel will measure pain at admission and discharge during the recovery phase.
Post-operative Pain | Measure at patient admission and discharge at 30 minute intervals.
  Pain scores will be measured through a reliable and validated observer-rated Children's Hospital of Eastern Ontario Pain Scale (CHEOPS) by two trained, blinded, and independent study personnel. Both study personnel will measure pain at admission and discharge during the recovery phase.

CONTACTS AND LOCATIONS:
Overall Officials: Luis Braga, MD, Principal Investigator — McMaster University
Locations (4):
- Canada (4):
  - McMaster Children's Hospital, Hamilton, Ontario
  - Children's Hospital, London Health Sciences Centre, London, Ontario
  - Children's Hospital of Eastern Ontario, Ottawa, Ontario
  - The Hospital for Sick Children, Toronto, Ontario